CLINICAL TRIAL: NCT00587899
Title: A Randomized, Single-blind Prophylactic Pulmonary Vein Isolation Procedure Utilizing Bipolar Radiofrequency Ablation in Patients Undergoing Mitral Valve Surgery
Brief Title: Prophylactic Pulmonary Vein Isolation Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment has been lower than anticipated due to growth in the minimally invasive mitral valve repair practice.
Sponsor: Mayo Clinic (Other)
Responsible Party: Thoralf, M. Sundt, III, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 06-005543
Record Dates: First submitted 2007-12-22; First posted 2008-01-08 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; AF; A fib; cardiac ablation; modified maze procedure
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): The treatment group will undergo operation for mitral valve disease with an additional procedure called Pulmonary Vein Isolation.
  Interventions: Procedure: Pulmonary Vein Isolation
- 2 (No Intervention): The control group of patients will undergo operation for mitral valve disease without the additional Pulmonary Vein Isolation

INTERVENTIONS:
Procedure: Pulmonary Vein Isolation — The treatment group will undergo operation for mitral valve disease with an additional procedure called Pulmonary Vein Isolation using a device that delivers radiofrequency energy to the heart muscle in order to create scar tissue to block electrical impulses that can trigger episodes of AF.
  Arms: 1

SUMMARY:
This study is being done to learn the effects of the Pulmonary Vein Isolation in patients that are at high risk to developing, but do not have a documented history of atrial fibrillation.

DETAILED DESCRIPTION:
Patients with a dilated left atrium (left upper chamber of the heart) that undergo mitral valve surgery may be at risk for the development of atrial fibrillation after surgery.

Atrial fibrillation (also known as "A-Fib" or AF) is an abnormal heart rhythm which may cause symptoms such as pounding sensations in your chest, dizziness, fatigue, chest pain and/or shortness of breath. AF patients are at a higher risk of developing a stroke.

Participants who sign informed consent will be randomized into one of two groups by chance (as in the flip of a coin).

Approximately 77 patients will undergo their mitral valve operation along with Pulmonary Vein Isolation (a treatment group) and 77 patients who do not undergo Pulmonary Vein Isolation at the time of their mitral valve surgery (a control group).

The treatment group will undergo operation for mitral valve disease with an additional procedure called Pulmonary Vein Isolation using a device that delivers radiofrequency energy to the heart muscle in order to create scar tissue to block electrical impulses that can trigger episodes of AF.

The control group of patients will undergo operation for mitral valve disease without the additional Pulmonary Vein Isolation.

ELIGIBILITY:
Inclusion Criteria:

* Indication for open-heart surgery: Mitral valve repair or replacement, evidence of a dilated left atrium

Exclusion Criteria:

* History of Atrial Fibrillation
* Need for emergent cardiac surgery
* Previous cardiac surgery
* Preoperative need for an intraaortic balloon pump or intravenous inotropes
* Current diagnosis of active endocarditis
* Mental impairment/or experience other conditions which may not allow subject to understand nature
* Significance and scope of study
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Evaluated by the number of patients free of taking antiarrhythmic medications and free of AF as determined by a 24-hour Holter recording. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Thoralf M. Sundt, III, M.D., Principal Investigator — Professor of Surgery, Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States